CLINICAL TRIAL: NCT03470194
Title: Urogynecological Office Visits and Patient Satisfaction of Limited English-Proficient Patients With Phone Interpreter Services Compared to In-Person Interpreters: Randomized Controlled Trial (SIPI)
Brief Title: Satisfaction of Limited English-Proficient Patients With Phone Interpretation Services Compared to In-Person Interpreters: A Randomized Controlled Trial
Acronym: SIPI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: H00013745
Record Dates: First submitted 2017-12-22; First posted 2018-03-19 (Actual); Results first posted 2021-04-05 (Actual); Last update posted 2021-04-05 (Actual); Status verified 2021-03

CONDITIONS: Pelvic Floor Disorders
Keywords: Quality Care; Access to health care; Interpretation services
MeSH Terms: conditions — Pelvic Floor Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interpretation Modality: In person (Active Comparator): Participants assigned to this group will use an in person interpreter for the duration of the UROGYN office visit
  Interventions: Other: Interpretation Modality: In Person
- Interpretation Modality: Telephonic (Active Comparator): Participants assigned to this group will use a phone interpreter for the duration of the UROGYN office visit
  Interventions: Other: Interpretation Modality: Telephonic

INTERVENTIONS:
Other: Interpretation Modality: In Person — Use of In-Person interpretation support for LEP participant during clinical appointment
  Arms: Interpretation Modality: In person
Other: Interpretation Modality: Telephonic — Use of telephonic interpretation support for LEP participant during clinical appointment
  Arms: Interpretation Modality: Telephonic

SUMMARY:
The aim of the study is to determine if In-person interpreters increases patient satisfaction of URGYN office visits compared to the use of phone interpreter services for Limited English Proficient (LEP) patients

DETAILED DESCRIPTION:
This study is a randomized controlled trial. Patients presenting to the UMass Memorial UROGYN clinic will be screened for eligibility using the inclusion and exclusion criteria. LEP patients will be identified as patients that initiate conversation in a non-English language and are only able to communicate adequately regarding their medical problem in a non-English language.

After patients have been seen for their scheduled office visit, they will be invited to participate in the study. Once the patient has agreed to participate in the study the participant will be randomized. Study assignment will be revealed using sequentially numbered sealed opaque envelopes. Randomization will be performed using software and a block randomization scheme to yield a 50% chance of having an in-person interpreter.

Those assigned to the control group will receive phone translation services and the experimental group will have in person interpreters.

At the subsequent visit, demographic information will be collected and patients will then receive interpretation services from the phone or an in-person interpreter.

ELIGIBILITY:
Inclusion Criteria:

* LEP speaking Spanish and Portuguese female patients presenting to the U Mass UROGYN clinic with or without Ad-hoc interpreters
* Spanish and Portuguese speaking female patients with LEP presenting to the U Mass UROGYN clinic for an office visit of any type

Exclusion Criteria:

* Unable to provide consent
* Under 18 years of age
* Pregnant women
* Prisoners
* LEP subjects who decline interpreter services
* Non -Spanish or Non - Portuguese speaking subjects
* Patients with cognitive impairment
* Visually or hearing impaired patients
* Patients not requiring a follow up appointment

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — female
Enrollment: 106 (Actual)
Dates: Start 2017-12-15 (Actual); Primary Completion 2019-06-10 (Actual); Study Completion 2019-06-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Flynn, MD, Principal Investigator — UMass Worcester
Locations (1):
- U Mass Memorial Hospital, Worcester, Massachusetts, United States

REFERENCES:
- [Derived] Taylor DL, Sierra T, Maheshwari D, Hall C, Leung K, Flynn M. Satisfaction With Telephone Versus In-Person Interpretation Services in Limited English-Proficient Urogynecology Patients: A Randomized Controlled Trial. Female Pelvic Med Reconstr Surg. 2021 Jun 1;27(6):388-392. doi: 10.1097/SPV.0000000000000880. PMID 32649326

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Interpretation Modality: In Person | Interpretation Modality: Telephonic
Started | 49 | 57
Completed | 38 | 40
Not Completed | 11 | 17
Not completed — Lost to Follow-up | 11 | 17

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Interpretation Modality: In Person | Interpretation Modality: Telephonic | Total
Number analyzed (Participants) | 49 | 57 | 106
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.3 (9.9) | 52.4 (13.8) | 54.1 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49 | 57 | 106
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 25 | 30 | 55
  Not Hispanic or Latino | 24 | 27 | 51
  Unknown or Not Reported | 0 | 0 | 0
Language of Translation [Count of Participants; unit: Participants]
  Spanish | 25 | 30 | 55
  Portugese | 24 | 27 | 51

OUTCOME MEASURES:

1. Primary Outcome: Patient Satisfaction
Description: Patient satisfaction will be measured by a 14 - item questionnaire. The questionnaire was created, validated, and used in a previous study from the field of Emergency medicine. There are 3 subscales assessing patient satisfaction with interpreter, nursing, and physician. Satisfaction with interpreters was calculated using the summation index of 4 items. Satisfaction with physician and nursing communication was measure by a summated index of 5 items that measure increasing level of satisfaction with a likert scale. Answers ranged from 1 to 4 where 4 equaled "strongly agree" and 1 equaled "strongly disagree". All items were weighted on a 100 point scale to facilitate interpretation of the means. A lower score means less satisfaction/greater dissatisfaction and a higher score indicates more satisfaction/less dissatisfaction.
Time Frame: Immediately assessed after office visit
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Interpretation Modality: In Person | Interpretation Modality: Telephonic
Number analyzed (Participants) | 38 | 40
score on a scale | 100 [92.9 to 100] | 94 [94.0 to 98.8]
Statistical Analysis 1: Comparison: Interpretation Modality: In Person vs Interpretation Modality: Telephonic; Test type: Other; p = 0.002, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: 1 week
Description: This did not involve any medical intervention which could result in a serious adverse event, mortality or other adverse events.
Arm/Group | Interpretation Modality: In Person | Interpretation Modality: Telephonic
All-Cause Mortality (participants affected / at risk) | 0/38 | 0/40
Serious Adverse Events (participants affected / at risk) | 0/38 | 0/40
Other Adverse Events (participants affected / at risk) | 0/38 | 0/40

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-10): https://cdn.clinicaltrials.gov/large-docs/94/NCT03470194/Prot_SAP_000.pdf